CLINICAL TRIAL: NCT06457243
Title: Closed-loop Neuromodulation Based on Individualised EEG Biomarkers of Methamphetamine Use Disorder
Brief Title: Closed-loop cTBS for the Core Clinical Features of Methamphetamine Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MZhao-019
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Amphetamine Use Disorders
Keywords: individualized therapy; closed-loop; Amphetamine-type stimulants; cTBS

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Closed-loop cTBS stimulation based on addiction-induced states (Experimental): In the initial phase of this study, participants will be subjected to individual closed-loop cTBS interventions at varying frequencies for one-week intervals. Concurrently, they will be exposed to MA-related cue paradigms to induce brain addiction states, while scalp EEG signals are collected. Stimulation will be initiated only upon identifying specific neural signals associated with MA cues, aiming to ascertain the optimal frequency for single-session closed-loop cTBS stimulation that could elicit individual neurological responses. Subsequently, we will embark on a longitudinal closed-loop cTBS intervention control study for MA dependents at one-week intervals, which involves addiction-induced closed-loop cTBS stimulation, random time-point stimulation, and traditional continuous stimulation, to rectify potential sequence effects and delineate the disparities in neurological and behavioral impacts between discrete and continuous stimulations based on brain states.
  Interventions: Device: Closed-loop cTBS stimulation based on addiction induced states

INTERVENTIONS:
Device: Closed-loop cTBS stimulation based on addiction induced states — We conducted a longitudinal controlled study of closed-loop cTBS interventions among MA dependents.This involved implementing interventions based on addiction-induced states through closed loop cTBS stimulation, randomized time-point stimulation, and traditional continuous stimulation.

SUMMARY:
Using specific EEG biomarkers in methamphetamine-dependent individuals, this study systematically probes closed-loop continuous Theta-burst Stimulation (cTBS) based on brain states, assessing dosage, neurologic and behavioral effects, while comparing its efficacy with traditional open-loop cTBS methods.

DETAILED DESCRIPTION:
The current study delineates a robust correlation between prefrontal cortex EEG signals and the psychological craving associated with methamphetamine usage. Dependents exhibit heightened β oscillation energy in the MPFC region and diminished γ oscillation energy across the DLPFC-MPFC region. Previously, through the implementation of rTMS interventions on the left DLPFC, the investigators have successfully reduced the craving levels in users when exposed to relevant cues, coupled with observed decreases in β oscillation energy and increases in γ oscillation energy in the MPFC region. This indicates that both β and γ oscillation energies are instrumental in representing the involvement of MPFC and DLPFC during craving episodes, and neuromodulatory technologies can modulate these energy levels, consequently reducing cravings. Furthermore, the investigators identified a significant augmentation in the theta energy in the occipital lobe when MA dependents are confronted with drug-related cue imagery, signifying a potential crucial neural marker for addiction-induced brain activity. Therefore, the investigators intend to employ the non-invasive continuous Theta-burst Stimulation (cTBS) , predicated upon biomarkers of addiction states, to administer specific frequency stimulations to targeted brain regions, aiming to achieve therapeutic objectives in addiction treatment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 60 years, irrespective of gender, having completed a minimum of 9 years of education and capable of effectively cooperating in questionnaire evaluations.
* Meet the diagnostic criteria set forth by the DSM-V concerning the amphetamine-type substance addiction.
* A history of utilizing amphetamine-type substances for a duration not less than one year, with a frequency of use being at least once per week.
* Consent to actively cooperate in the completion of subsequent follow-up assessments.

Exclusion Criteria:

* Severe cognitive functional impairments manifested through a history of head trauma, cerebrovascular diseases, epilepsy, etc., or usage of cognitive enhancement drugs in the past 6 months; an intellectual disability with an IQ score less than 70.
* A diagnosis of schizophrenia or other severe mental illnesses as per the DSM-5 criteria.
* Abuse or dependence on other psychoactive substances (excluding nicotine) within the past 5 years.
* Severe organic diseases that might compromise study participation.
* Contraindications to cTBS, such as a history of epileptic seizures or the presence of metallic implants in proximity to the head.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change of Craving assessed by Visual Analog Scale (VAS) | through study completion, an average of 1 month
  The intensity of psychological craving in MA dependents was assessed using the Visual Analogue Scale (VAS), where individuals rated their cravings on a scale from 0 to 10, with higher scores indicating greater levels of craving. The VAS scores were utilized based on two conditions: during a resting state and when subjected to cue induction involving images associated with methamphetamine, serving as the criteria for evaluation.
  individuals rated their cravings on a scale from 0 to 10, with higher scores indicating greater levels of craving. The VAS scores were utilized based on two conditions: during a resting state and when subjected to cue induction involving images associated with methamphetamine, serving as the criteria for evaluation.

SECONDARY OUTCOMES:
Changes of electroencephalogram power spectrum | through study completion, an average of 1 month
  Resting-state EEG can be used to extract power spectra and electrode functional connectivity; on-task EEG can be used to isolate time-frequency features during non-stimulated trials to extract alpha, beta, theta, and gamma band energy of the parietal and occipital electrodes. Both can be used to assess changes in neural activity before, during, and after their restimulation.
Probabilistic inversion learning task | through study completion, an average of 1 month
  The matching of symbols and colours was reversed without informing the subjects and their cognitive flexibility in the reversed condition was assessed
Anxiety | through study completion, an average of 1 month
  The reduction rate in the Beck Anxiety Inventory (BAI) scores was calculated before and after intervention to assess the rate of decrease in anxiety levels among MA dependents.
Depression | through study completion, an average of 1 month
  The reduction rate in the Beck Depression Inventory (BDI) scores was calculated before and after the intervention to evaluate the rate of reduction in their levels of depression.
sleep quality | through study completion, an average of 1 month
  Improvement in subjects' sleep before and after the intervention as assessed by the Pittsburgh Sleep Quality Index scale (PSQI)

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhao, PhD, Study Chair — Shanghai Mental Health Center
Locations (1):
- Min Zhao, PhD, Shanghai, Shanghai Municipality, China